CLINICAL TRIAL: NCT02649868
Title: A Phase II Study Using LC Bead LUMI Radio-Opaque Embolic Beads to Detect and Characterize the Vascularity of Hepatic Tumors During Treatment With Transarterial Embolization (TAE) Alone or Combined With Thermal Ablation
Brief Title: LC Bead LUMI Radio-Opaque Embolic Beads to Detect and Characterize the Vascularity of Hepatic Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailability of study device
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 160049; 16-CC-0049
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Cancer; Liver Neoplasms; Hepatocellular Cancer; Liver Cancer
Keywords: Radio-Opaque Bland Beads; Thermal Ablation; Transarterial Embolization
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hepatic tumors bead embolization (Experimental): Participants with diagnosed hepatic malignancy underwent transarterial embolization (TAE) with or without thermal ablation under general anesthesia. The LC LUMI bead were used in the transarterial embolization procedure.
  Interventions: Procedure: Transarterial embolization (TAE); Device: LC Bead LUMI

INTERVENTIONS:
Procedure: Transarterial embolization (TAE) — Transarterial embolization
Device: LC Bead LUMI — LC Bead LUMI has been designed as a radiopaque version of the LC Bead

SUMMARY:
Background:

Liver cancer begins in the cells of the liver. It can be treated with chemotherapy, radiation, or even a liver transplant. A less invasive treatment may be able to help some people with liver cancer. It is called percutaneous transarterial embolization (TAE). For TAE, a material is injected into blood vessels to block the blood flow that is feeding the tumor. Researchers want to test a new material for TAE that may shrink tumors and can be seen on x-ray and CT images. The embolization may sometimes be combined with thermal ablation, or cooking tumors with needles that deliver heat by electricity or microwave.

Objective:

To test an embolization material called an LC LUMI beads. To see if it can block blood vessels that provide blood to cancerous tumors and to see how the beads look on x-ray and CT images.

Eligibility:

Adults 18-85 years old who have been diagnosed with liver cancer

Design:

Participants will have routine blood tests, physical exams, and x-rays.

Participants will be screened with blood tests, physical exam, and medical history. They will have a computed tomography (CT) scan of the abdomen and pelvis. This will include a contrast drink and a contrast (dye) injected in the veins.

Participants will be admitted to the clinic. They will repeat the screening tests.

Participants may have other tests. These may include x-rays, other scans, or ultrasound.

Participants will be evaluated for general anesthesia.

They will get counseling about the procedure.

Participants will get anesthesia. The LC LUMI beads will be injected into blood vessels. The beads contain iodine, which makes them visible by x-ray and by a CT scan machine.

Participants will have follow-up visits for 12 months. They will have CT scans and/or other radiologic tests.

DETAILED DESCRIPTION:
Background:

Hepatocellular Carcinoma (HCC) is the 3rd most common cause of cancer globally with an increasing incidence worldwide.

Management of hepatic malignancies from primary Hepatocellular Carcinoma (HCC) or metastatic disease involves a multidisciplinary approach of surgery and chemotherapy and in the case of HCC, transplant, anti-VEGF sorafenib, or local or regional image guided therapies.

Thermal ablation (RFA or MWA) and transarterial embolization (TAE) are minimally invasive image guided local or regional therapies that have been extensively studied for decades, and more recently and to a lesser extent have been studied together as a combination therapy.

LC Bead LUM^TM, a radiopaque embolic bead product (company code BTG 13-002), is an imageable spherical embolic product that can be visualised by X-ray based imaging (e.g., fluoroscopy and CT).

The beads are non-resorbable microspheres with calibrated size ranges that occlude arteries for the purpose of blocking the blood flow to a target tissue.

LC Bead LUMITM are intended to be used for the embolization of hypervascular tumors and arteriovenous malformations (AVMs).

Objectives:

To determine the imaging characteristics of radiopaque beads including qualitatively comparing virtual and actual bead perfusion in the treatment of hepatic tumors using bead embolization.

Eligibility:

Treatment eligibility for TAE requires agreement between the Interventional Radiologist reviewing imaging and feasibility of TAE and the patient's NIH primary treatment team who will evaluate the patient's clinical parameters to undergo anesthesia and the TAE and or ablation procedure.

At least >=18 years of age

Patients with pathologically proven, hepatic-dominant neoplasm.

The extent of hepatic metastases is <50% of total hepatic volume.

Past treatment with Y90 must be 6 months from TAE treatment and liver function within NIH institutional limits

ECOG performance status <=2

Patients must have normal organ and marrow function per laboratory parameters

Patients with minor allergies to iodine will also be excluded.

Design:

Number of Participants: 30

Recruitment Time Frame: approximately 2 years

Type of Study: Feasibility study

This is a pilot study to assess the characteristics of radio-opaque bland beads during TAE in the treatment of hepatic malignancies. Patients may also receive thermal ablation treatment in conjunction with TAE if clinically indicated, although comparison of bead treatment with or without thermal ablation is not part of the study s aim.

To compare virtual and actual perfusion characteristics of the LUMI radiopaque beads with CBCT and/or CT. Patients scans will be obtained per TAE standard of care schedule. Other imaging evaluation of this therapy may be performed at regular intervals following completion of treatment, and will be governed by standard conventional imaging regimen post treatment.

The choice of which combination of imaging (CT, Cone beam CT (CBCT), or fluoroscopy) and when to image, will be made by the clinical care team for the patient, based upon multidisciplinary recommendations and NIH Clinical Center customary use and standard of care, and will be purely clinical decisions (not research-related).

The participants will have a diagnosed hepatic malignancy, and be eligible to undergo transarterial embolization and thermal ablation under general anesthesia. The LC LUMI bead will be used in the transarterial embolization procedure.

Follow up will continue for 12 months from the time of initial treatment.

Patients will be evaluated in multidisciplinary GI medical oncology clinic and up to 30 patients will be enrolled to accrue 20 evaluable patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients who are determined to be eligible for TAE by an interventional radiologist and the primary/referring team will be eligible for the study.
* Patients with pathologically proven hepatic-dominant neoplasm that might otherwise be candidates for standard clinical TAE.
* Extent of hepatic metastases is <50% of total hepatic volume.
* At least >=18 years of age: Because it is exceeding rare for someone under the age of 18 to develop hepatocellular carcinoma, we will exclude patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status 0-2
* Six months since last treatment with Y90
* Patients must have normal or adequate organ and marrow function as defined below:

  * Hematology/Absolute Neutrophil Count/ > 1500 / mm^3 without help of Filgrastim or other stimulating growth factors
  * Hematology/Platelet Count Patient eligible if platelet count is correctable to >=50,000/mm^3
  * Hematology/Hemoglobin Patient eligible if hemoglobin count is correctable to >= 8.0 g/dl
  * Serum Chemistry/ALT/AST <= 5 times the upper limit of normal; except in the presence of obstructive liver metastases where ALT/AST may be up to 10 times the upper limit of normal
  * Serum Chemistry/Creatinine <1.5x institution upper limit of normal OR creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
  * Serum Chemistry/Total Bilirubin <=3 mg/dl
  * Serum Chemistry/Prothrombin Time within 2 seconds of the upper limit of normal (INR<=1.8)
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

EXCLUSION CRITERIA:

* No contraindications to receive iodine products.
* Main Portal Vein Occlusion or other contraindications to chemoembolization
* Patients taking immunosuppressive drugs or unable to come off of ongoing chronic anticoagulation will not be eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection with systemic manifestations, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and nursing mothers are excluded from this study because of the potential for teratogenic or abortifacient effects of required multiple imaging and associated radiation doses, anesthesia and risks during thermal ablation to the fetus. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford J Wood, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.Plan to share human data generated in this research for future research as follows:
  * De-identified data in BTRIS
  * De-identified or identified data with approved outside collaborators under appropriate agreements
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the time of publication or shortly thereafter
Access Criteria: De-identified data in Biomedical Translational Research Information System (BTRIS)
  De-identified or identified data with approved outside collaborators under appropriate agreements

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0049.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 19 participants who were consented, two participants were unevaluable so were excluded from the study
Period: Overall Study
Arm/Group | Hepatic Tumors Bead Embolization
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hepatic Tumors Bead Embolization
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Perfusion Characteristics of Imageable Beads Using Cone Beam CT
Description: Perfusion on x-ray was assessed after delivery of transarterial embolization beads. Qualitative geometric analysis of actual and virtual perfusion was performed with data available using custom software analysis after selective injections of image-able beads during transcatheter intra-arterial delivery to the liver. Liver boundary and super selective perfused boundary were segmented and compared for distribution of beads on virtual and actual perfusion for possible match. Analysis was the visibility of beads upon transcatheter intra-arterial delivery to the liver and evaluation of impact on perfusion from subjective evaluation during procedural angiography, and/or cone beam CT. Qualitative analysis was done to determine match for distribution of beads on virtual and actual perfusion.
Time Frame: Intra-procedure
Population: Participants who completed the transcatheter intra-arterial (TAE) procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatic Tumors Bead Embolization
Number analyzed (Participants) | 17
Participants
  Yes | 17
  No | 0

2. Primary Outcome: Perfusion Characteristics of Imageable Beads Using Cone Beam CT
Description: as for outcome 1
Time Frame: One year post procedure
Population: Participants who completed the transcatheter intra-arterial (TAE) procedure and had one year follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatic Tumors Bead Embolization
Number analyzed (Participants) | 12
Participants
  Yes | 12
  No | 0

ADVERSE EVENTS:
Time Frame: Up to one year post procedure
Arm/Group | Hepatic Tumors Bead Embolization
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatic Tumors Bead Embolization (N=17)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Edema peripheral (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Subdural haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatic Tumors Bead Embolization (N=17)
Anemia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Chest pain (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastroparesis postoperative (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 5
Administration site lymphadenopathy (General disorders) | 1
Asthenia (General disorders) | 1
Axillary pain (General disorders) | 1
Chills (General disorders) | 2
Edema peripheral (General disorders) | 4
Face edema (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 7
Flank pain (General disorders) | 3
Flushing (General disorders) | 2
Hyperthermia (General disorders) | 12
Hypothermia (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Night sweats (General disorders) | 1
Pain (General disorders) | 9
Pelvic mass (General disorders) | 1
Biloma (Hepatobiliary disorders) | 1
Medical device site bruise (Injury, poisoning and procedural complications) | 1
Absolute neutrophil count decreased (Investigations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 7
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 4
Blood lactate dehydrogenase (Investigations) | 1
International normalized ratio increased (Investigations) | 1
Platelet count decreased (Investigations) | 5
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 2
Anorexia nervosa (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7
Groin pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Confusional state (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 9
Insomnia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Micturition urgency (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Urinary tract infection (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2
Paralysis recurrent laryngeal nerve (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin papilloma (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 1
Portal vein thrombosis (Vascular disorders) | 1
Procedural haemorrhage (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT02649868/Prot_SAP_000.pdf